CLINICAL TRIAL: NCT06697028
Title: Assessment of Cardiorespiratory Fitness Using the Progressive Aerobic Cardiovascular Endurance Run in Patients With Juvenile Idiopathic Arthritis and Familial Mediterranean Fever: A Healthy Control Study
Brief Title: Assessment of Cardiorespiratory Fitness Using the PACER in Patients With Juvenile Idiopathic Arthritis and Familial Mediterranean Fever
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Asya Albayrak, MSc, Istanbul Kent University
Other Study IDs: AAlbayrak
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-12

CONDITIONS: Juvenile Idiopathic Arthritis; Familial Mediterranean Fever; Healty Controls
Keywords: Cardiorespiratory fitness; Progressive Aerobic Cardiovascular Endurance Run; Body composition; Maximum oxygen consumption; Juvenile Idiopathic Arthritis; Familial Mediterranean Fever
MeSH Terms: conditions — Arthritis, Juvenile; Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Juvenile Idiopathic Arthritis: Patients diagnosed with JIA followed at the Pediatric Rheumatology Clinic, Department of Pediatrics, Istanbul Faculty of Medicine, will be evaluated.
  Interventions: Other: Usability and Comparison
- Familial Mediterranean Fever: Patients diagnosed with FMF followed at the Pediatric Rheumatology Clinic, Department of Pediatrics, Istanbul Faculty of Medicine, will be evaluated.
  Interventions: Other: Usability and Comparison
- Healthy control: The outcomes of individuals with rheumatic diseases will be compared with those of healthy controls.
  Interventions: Other: Usability and Comparison

INTERVENTIONS:
Other: Usability and Comparison — PACER will be used to assess cardiorespiratory fitness in individuals with rheumatic diseases. The results will be compared with those of healthy individuals, and the relationship between body composition and VO2 max will be examined.

SUMMARY:
Juvenile Idiopathic Arthritis (JIA) and Familial Mediterranean Fever (FMF) are the most common autoimmune and autoinflammatory rheumatic diseases in childhood. Symptoms such as reduced muscle strength, joint pain, fatigue, and limited activity, which are common in childhood rheumatic diseases, often lead to impaired physical function. Cardiorespiratory fitness, which is an important indicator of physical function, plays a critical role in health-related outcomes in children and adolescents with rheumatic disease. Maximum oxygen consumption (VO2 peak) is considered the fundamental criterion for evaluating cardiorespiratory fitness. The need for extensive equipment and trained personnel, accompanied with the inability to assess large numbers of children at one-time makes the objective assessment of cardiorespiratory fitness in a clinic setting unmanageable. Therefore, there is a need to assess their cardiorespiratory fitness utilizing an easily administered test that has minimal measurement errors in patients with JIA and FMF. The Progressive Aerobic Cardiovascular Endurance Run (PACER) has become a routine cardiorespiratory fitness assessment for predicting VO2peak in children. A review of the literature revealed that no studies have evaluated CRF using PACER in childhood rheumatic diseases. The aim of this study was to compare the Fitnessgram VO2 max values of children and adolescents diagnosed with JIA and FMF with those of their healthy peers and to examine the relationship with body composition.

ELIGIBILITY:
Inclusion Criteria:

* Did not have any chronic disease other than rheumatic disease
* Diagnosed with rheumatic disease at least 6 months ago
* Had stable medical treatment
* Being between the ages of 12 and 18
* Volunteering to participate in the study

Exclusion Criteria:

* Have experienced trauma or surgery affecting the musculoskeletal system within the last 6 months
* Have acute pain for any reason, have visual or hearing problems
* Have cognitive impairment
* Not volunteering to participate in the study

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients diagnosed with JIA and FMF, and their healthy peers without any chronic diseases or disabilities, all aged between 12 to 18 years old will be evaluated with PACER.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-01-11 (Actual); Study Completion 2025-05-11 (Actual)

PRIMARY OUTCOMES:
Progressive Aerobic Cardiovascular Endurance Run (PACER) | Baseline
  The PACER test is an adapted version of the 20-meter shuttle run test and consists of multiple stages, serving as a field test. It allows children and adolescents to set their own pace and warm up, serving as a more enjoyable alternative to other distance running tests recommended for use in children, adolescents, and young adults. Utilized to assess patients' cardiorespiratory fitness, individuals were instructed to run back and forth between two cones within a 20-meter course, to the rhythm of music played through a sound recording device, with the test starting at a slow pace and gradually increasing in speed every minute.
Body Mass Index | Baseline
  Body mass index (BMI), will determined by dividing the body weight in kilograms by the square of the height in meters.
VO2 max | Baseline
  Using the FitnessGram software, the maximum oxygen consumption value (VO2max) will calculated for each individual based on the number of laps completed.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No